CLINICAL TRIAL: NCT02712463
Title: A Retrospective, Observational Study to Assess the Rate of Hospitalization in Patients With Schizophrenia Treated One Year Before With Oral Antipsychotics and One Year After With Long Acting Injectable Atypical Antipsychotics - REALAI Study
Brief Title: A Study to Assess the Rate of Hospitalization in Participants With Schizophrenia Treated With Antipsychotics
Acronym: REALAI
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107059; R092670SCH4039 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Oral antipsychotics; Long acting Injectable antipsychotics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Schizophrenia: This is an observational study. Data will be collected from the medical records of participants diagnosed with schizophrenia and who had been on oral antipsychotics for at least one year and thereafter have been switched to Long Acting Injectable atypical antipsychotics for at least one year.

SUMMARY:
The primary purpose of the study is to compare the rate of hospitalization associated with psychotic relapse in participants with schizophrenia treated one year before with oral antipsychotics and one year after with long acting injectable atypical antipsychotics.

DETAILED DESCRIPTION:
This is a retrospective (take a look back at events that already have taken place), observational, multicenter (when more than one hospital or medical school team work on a medical research study) study to review medical records of adults with a diagnosis of Schizophrenia during the time period from 01 January 2009 through 31-December-2013 (only for Mexican population). Data will be collected from clinical practice. The medical records of participants will be screened and eligible participants data will be collected. The period of observation will span from 12 months before initial Long Acting Injectable (LAI) use and in 12 months after the initial LAIs use. The rate of hospitalization will be primarily evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Out-Patients with the main diagnosis of schizophrenia with Diagnostic and Statistical Manual of Mental Disorders (DSM-4 criteria)
* Only clinical records with complete information during the 2 years period selected for data analysis will be included
* Participants treated with oral antipsychotics then switched to Long Acting Injectable (LAI) due to poor adherence, lack of efficacy (no significant symptom reduction, judged by physician, at maximum recommended dose of an antipsychotic for 6 weeks), or participants choice, (Excluding for the Brazil population, when the switch has not been clearly justified or the switch has not been done during hospitalization)
* Being regularly treated with LAI atypical antipsychotics for at least 1 year after the initial use of LAI atypical antipsychotics

Exclusion Criteria:

* Participants with refractory schizophrenia (RS)
* Participants that started LAI treatment as in-patients and patients that switched to LAI during hospitalization (only for Mexican population).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants (both gender and 18 to 55 years of age) with schizophrenia treated with oral anti-psychotics then switched to long acting Injectable anti-psychotics.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Hospitalizations in 12 Months Before Initial Long Acting Injectable anti-psychotics (LAI) use | 12 months before initial LAI use
  Percentage of participants with hospitalizations due to Psychotic relapse of schizophrenia will be reported.
Percentage of Participants with Hospitalizations in 12 Months After Initial Long Acting Injectable anti-psychotics (LAI) use | 12 months after initial LAI use

SECONDARY OUTCOMES:
Number of hospitalizations due to Psychotic Relapse of Schizophrenia | approximately 2 years
  The number of hospitalizations due to Psychotic relapse of schizophrenia will be reported.
Number of Days of Hospitalization due to Psychotic Relapse of Schizophrenia | approximately 2 years
  The number of days of hospitalization due to Psychotic relapse of schizophrenia will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (11):
- Brazil (5):
  - Aracaju
  - Brasília
  - Rio de Janeiro
  - São José
  - São Paulo
- Mexico (6):
  - Durango
  - Hermosillo
  - Ixtapaluca
  - México
  - Monterrey
  - San Pedro Garza García